CLINICAL TRIAL: NCT01742299
Title: An Open Label, Multi-center Imatinib Roll-over Protocol for Patients Who Have Completed a Previous Novartis-sponsored Imatinib Study and Are Judged by the Investigator to Benefit From Continued Imatinib Treatment
Brief Title: Study to Allow Access to Imatinib for Patients Who Are on Imatinib Treatment in a Novartis-sponsored Study and Are Benefiting From the Treatment as Judged by the Investigator
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571A2406; 2012-002540-25 (EudraCT Number)
Record Dates: First submitted 2012-11-28; First posted 2012-12-05 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: GIST and CML
Keywords: Glivec/Gleevec; CML; GIST; Imatinib mesylate
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- imatinib mesylate (Experimental): The starting dose of imatinib should be the same as the last dose that was given in the parent imatinib study (400 mg/day to 600 mg/day). After this, the dose of imatinib is based on the investigator's judgment.
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate — Imatinib will be provided as 100 mg and 400 mg tablets taken orally once daily unless other wise instructed by investigator
  Other Names: STI571

SUMMARY:
The purpose of this study is to allow continued use of imatinib in patients who are on imatinib treatment in a Novartis-sponsored, Oncology Clinical Development & Medical Affairs (CD&MA) study and are benefiting from the treatment as judged by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is currently enrolled in a Novartis-sponsored, Oncology Clinical Development & Medical Affairs study receiving imatinib and has fulfilled all their requirements in the parent study. 2.Patient is currently benefiting from the treatment with imatinib, as determined by the investigator. 3. Patient has demonstrated compliance, as assessed by the investigator, with the parent study protocol requirements.4. Willingness and ability to comply with scheduled visits, treatment plans and any other study procedures. 5. Written informed consent obtained prior to enrolling in roll-over study. 6.If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.

   Exclusion Criteria:
   * 1. Patient has been permanently discontinued from imatinib treatment in the parent study due to unacceptable toxicity, non-compliance to study procedures, withdrawal of consent or any other reason.
2. Patient has participated in a Novartis sponsored combination trial where imatinib was dispensed in combination with another study medication and patient is still receiving combination therapy.
3. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hcG laboratory test.
4. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during the study and for 30 days after the final dose of imatinib. Male patients must use highly effective contraception during the study and for 30 days after the final dose of imatinib.

Highly effective contraception is defined as either:

* Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* Male sterilization (at least 6 months prior to enrolling). For female patients on the study the vasectomized male partner should be the sole partner for that patient.
* Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.

In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

If a study patient becomes pregnant or suspects they are pregnant during the study or within 30 days of the final dose of imatinib, the Investigator/Study Doctor needs to be informed immediately and ongoing study treatment with imatinib has to be stopped immediately.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2013-03-26 (Actual); Primary Completion 2033-04-21 (Estimated); Study Completion 2033-04-21 (Estimated)

PRIMARY OUTCOMES:
To evaluate long term safety data (SAEs and AEs) | Until no patients are left on study, with an expected average of 20 years
  To better characterize the long-term safety of imatinib in patients who are on imatinib treatment and are benefiting from the treatment as judged by the investigator

SECONDARY OUTCOMES:
To evaluate clinical benefit as assessed by the investigator. | Until no patients are left on study, with an expected average of 20 years
  To better characterize the long-term safety of imatinib in patients who are on imatinib treatment and are benefiting from the treatment as judged by the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (26):
- United States (9):
  - University of California LA, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - Sidney Kimmel CCC At JH, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Weill Cornell Medical Center, New York, New York
  - Oregon Health Sciences University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Uni Of TX MD Anderson Cancer Cntr, Houston, Texas
- China (4):
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Helsinki, Finland
- France (3):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Poitiers
- Novartis Investigative Site, Hong Kong, Hong Kong
- Romania (2):
  - Novartis Investigative Site, Cluj-Napoca, Cluj
  - Novartis Investigative Site, Bucharest
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Basel, Switzerland
- Novartis Investigative Site, Bangkok, Thailand
- Novartis Investigative Site, Ankara, Sihhiye-Altindag, Turkey (Türkiye)
- United Kingdom (2):
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com